CLINICAL TRIAL: NCT02963753
Title: Effect of Hyperemesis Gravidarum on 75 Gram Oral Glucose Tolerance Test Screening and Gestational Diabetes Mellitus
Brief Title: Hyperemesis Gravidarum and 75 Gram Oral Glucose Tolerance Test
Status: Completed | Type: Observational
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf MADENDAG, Principal Investigator, Kayseri Education and Research Hospital
Other Study IDs: 2017/173
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Hyperemesis; Gravidarum, With Dehydration; Gestational Diabetes
Keywords: Hyperemesis gravidarum; gestational diabetes mellitus; oral glucose tolerance test
MeSH Terms: conditions — Hyperemesis Gravidarum; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- hyperemesis gravidarum group: The study group consisted of women hospitalized for hyperemesis during first trimester of their pregnancy
- the control group: whereas the control group included all other women who delivered in the same period.

SUMMARY:
Hyperemesis gravidarum (HEG) is not only nausea and vomiting of pregnancy, but it is also a clinical syndrome including endocrine and metabolic complications. Recently, some investigators have been begun performing researches related to the development of gestational diabetes mellitus (GDM) in pregnant women with HEG because they think about those metabolic and endocrine complications of HEG.In the literature there are few studies assessing how HEG has effects on GDM or 75 gram oral glucose tolerance test (OGTT). So the investigators aim to evaluate the effects of HEG on 75 gram OGTT.

DETAILED DESCRIPTION:
This retrospective controlled study conducted by Obstetrics and Gynecology clinics of Kayseri Training and Research Hospital.Pregnant women who delivered at the Kayseri Education and Training Hospital of Medicine, in Turkey, between January 2010 and September 2016 were identified.This study was carried out with two groups. The study group consisted of women hospitalized for Hyperemesis gravidarum (HEG) during first trimester of their pregnancy, whereas the control group included all other women who delivered in the same period.Screening for GDM was performed twice during pregnancy. The first screening was performed during the first trimester using the random plasma glucose test with a cutoff value of 109 mg/dl. Screening for GDM was performed for all women during their first prenatal visit, regardless of the presence or absence of hyperemesis-associated symptoms.The second screening was performed during the second trimester, between 24 and 27 weeks, using a 75-g oral glucose tolerance test (OGTT), after pregnant women with HEG got rid of hyperemesis. GDM was diagnosed on the basis of the universal criteria established by the International Association of Diabetes and Pregnancy Study Group: a plasma glucose level that met or exceeded the fasting cutoff value 92 mg/dl, the first-hour cutoff value 180 mg/dl, or the second-hour cutoff value 153mg/dl.

To be considered for diagnosis of pre-gestational diabetes mellitus, women had to meet at least one of the following criteria: the fasting plasma glucose test with a cutoff value of 126 mg/dl or the random plasma glucose test with a cutoff value of 200 mg/dl or the second-hour cutoff value 153mg/dl after 75 gram OGGT (American Diabetes Association) The delivery midwifery and medical records were retrospectively evaluated. All of the patient's body mass index (BMI,calculated as weight in kilograms divided by the square of height in meters), urine ketone levels and ages were recorded separately both in the initial exam and during performing 75 gram OGTT.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 35 years-old singleton pregnancies and performed 75 gram OGTT

Exclusion Criteria:

* Other causes lead to nausea and vomiting in pregnancy such as gastroenteritis, gastroparesis, hepatitis, intestinal obstruction, peptic ulcer, appendicitis, pyelonephritis, urolithiasis, ovarian torsion, diabetes mellitus, hyperthyroidism, hyperparathyroidism, migraine.
* And also patients who have risks for GDM such as body mass index > 30, history of GDM in previous pregnancy and diabetes in the family were excluded.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study was carried out with two groups. The study group consisted of women hospitalized for HEG during first trimester of their pregnancy, whereas the control group included all other women who delivered in the same period. When the pregnant women had those symptoms such as the presence of intractable vomiting during pregnancy associated with dehydration, electrolyte,and/or metabolic disturbances, as well as a weight loss 5% or more, they were diagnosed as HEG.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
To determine serum glucose levels in both groups during 75 gram oral glucose tolerance test screening | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: YUSUF MADENDAG, Principal Investigator — Kayseri Education and Research Hospital